CLINICAL TRIAL: NCT01462877
Title: An Open-label, Multi-center Study to Evaluate the Efficacy and Safety of Statin-fenofibrate Combination Therapy in Dyslipidemic Chinese Patients
Brief Title: A Study to Evaluate Fenofibrate Combination With Statin in Chinese Patients With Dyslipidemic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Rundo International Pharmaceutical Research & Development Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W13-254
Record Dates: First submitted 2011-10-28; First posted 2011-11-01 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Dyslipidemias; Cardiovascular Diseases; Hypertriglyceridemia
Keywords: Lipid Regulating Agents; Drug Therapy; cardiovascular diseases; hypertriglyceridemia; Hydroxymethylglutaryl-CoA Reductase Inhibitors; fenofibrate; Dyslipidemias; Combination
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases; Hypertriglyceridemia | interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fenofibrate arm (Other)
  Interventions: Drug: fenofibrate

INTERVENTIONS:
Drug: fenofibrate — Fenofibrate Capsule 200mg qd orally
  Other Names: ABT-799; lipanthyl

SUMMARY:
Atherogenic dyslipidemia includes patients who have coronary heart disease (CHD) or CHD risk equivalents, whose TG level is not adequately controlled after statin monotherapy. According to the published ESC/EAS consensus, fibrate is suggested to be added to this type of patient who has insufficient improvement. The purpose of the study is to evaluate the efficacy on lipid control and the safety of adding fenofibrate in patients on a background of statin treatment.

DETAILED DESCRIPTION:
It is an open-label , single group, multi-center study. At around 30 investigate sites, 500 dyslipidemic Chinese patients with coronary heart disease (CHD) or CHD risk equivalent, whose TG ≥1.70 mmol/L (150mg/dl) and <5.65mmol/L (500mg/dl) after at least 2 month statin monotherapy with standard dose will be enrolled. After at least 2 month statin monotherapy with standard dose, patients having high TG will be recruited and given statin-fenofibrate combination therapy for 8 weeks. Several lipid parameters and safety parameters will be compared between baseline, after 4 weeks treatment and after 8 weeks treatment. Primary efficacy endpoint is the percentage of TG decrease before and after 8 weeks treatment. Secondary endpoints on efficacy are the absolute change and the percent of change on TC, LDL-C, HDL-C, apoA1, apoB and apoB/apoA1 of baseline, after 4 weeks treatment and 8 weeks treatment, absolute change and percentage of change of hsCRP from baseline to 8 weeks of treatment. Second endpoints on safety is the incidence of AE/SAE, change on CK, ALT, AST, BUN and Cr before and after treatment and the number of clinical meaningful abnormal change defined as ALT or AST >3ULN, or CK >10ULN, or BUN >1.5ULN or Cr >1.5ULN. Other Arm type is a self comparator

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years and < 80 years, male or female
2. With at least one risk of coronary heart disease (CHD) [medical history of myocardial infarction (MI) or coronary angiography shows coronary stenosis ≥ 50% or post percutaneous coronary intervention (PCI) or post coronary artery bypass grafting (CABG)] or CHD risk equivalents, which comprise,

   * Other clinical forms of atherosclerotic disease (ischemic stroke, peripheral arterial disease, abdominal aortic aneurysm, and symptomatic carotid artery disease)
   * Type 2 Diabetes
   * Multiple risk factors that confer a 10-year risk for CHD >20%.
3. ≥ 2 months statin monotherapy with standard dose (atorvastatin ≤20mg q.d. or rosuvastatin ≤10mg q.d. or simvastatin ≤40mg q.d. or pravastatin ≤40mg q.d. or pitavastatin ≤4mg q.d or fluvastatin ≤80mg q.d. or lovastatin ≤40mg q.d.) and plan to continue the previous type and dose of statin
4. Triglycerides (TG)≥1.70 mmol/L (150mg/dl) and TG<5.65 mmol/L (500mg/dl)
5. Subject must be able to provide informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), on his or her own behalf, prior to any study-specific procedures.

Exclusion Criteria:

1. Hypersensitive to fenofibrate or to any of its excipients
2. Hepatic insufficiency [alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2ULN (upper limit of normal)]
3. Renal insufficiency [Creatinine clearance rate (Ccr)<60ml/min estimated from Cockcroft-Gault equation Ccr=(140-age)*weight(Kg)*0.85(if female)/[0.818*Cr (µmol/L)]
4. Creatine kinase (CK) > 2 ULN
5. Congenital galactosemia, glucose-galactose malabsorption syndrome or lactase deficiency
6. Hypothyroidism
7. Combination use of other non-statin lipid-regulating drugs such as fibrates, niacin and fish oil in previous 2 months
8. Combination use of drug with similar structure as Fenofibrate, especially ketoprofen
9. Combination use of oral anticoagulants
10. Pregnant or lactating woman
11. Other conditions at investigator's discretion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyra Xie, MD, Study Chair — Abbott
Locations (1):
- Site Reference ID/Investigator# 64695, Xiamen, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dyslipidemic Chinese patients with CHD or CHD equivalent, whose TG ≥1.70 mmol/L and <5.65mmol/L after at least 2 month statin monotherapy with standard dose were enrolled. After at least 2 month statin monotherapy with standard dose, patients having high TG were recruited and given statin-fenofibrate combination therapy for 8 weeks.
Period: Overall Study
Arm/Group | Fenofibrate Arm
Started | 506
Safety Set | 492
Full Analysis Set | 468
Per-protocol Set | 364
Completed | 435
Not Completed | 71

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 468
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194
  Male | 274
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 130.93 (12.50)
diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 78.54 (8.97)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Triglyceride (TG) Change
Description: Blood tests
Time Frame: Baseline and up to 8 weeks after intervention
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of TG change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 468
percentage of TG change | -38.12 (33.92)

2. Secondary Outcome: Change in Serum Total Cholesterol
Description: Blood tests
Time Frame: Baseline and up to 8 weeks after intervention
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of TC change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 468
percentage of TC change | 2.75 (24.75)

3. Secondary Outcome: Change in Serum Low-density Lipoprotein Cholesterol
Description: Blood tests
Time Frame: Baseline up to 8 weeks after intervention
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of LDL-C change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 468
percentage of LDL-C change | 14.91 (39.80)

4. Secondary Outcome: Change in Serum High-density Lipoprotein Cholesterol
Description: Blood tests
Time Frame: Baseline up to 8 weeks after intervention
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of HDL-C change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 468
percentage of HDL-C change | 17.40 (32.62)

5. Secondary Outcome: Change in Serum Non-high-density Lipoprotein Cholesterol
Description: Blood tests
Time Frame: Baseline up to 8 weeks after intervention
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of Non-HDL-C change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 468
percentage of Non-HDL-C change | -1.30 (28.26)

6. Secondary Outcome: Change in Serum Apolipoprotein A1
Description: Blood tests
Time Frame: Baseline up to 8 weeks after intervention
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of apoA1 change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 468
percentage of apoA1 change | 12.41 (28.74)

7. Secondary Outcome: Change in Serum Apolipoprotein B
Description: Blood tests
Time Frame: Baseline up to 8 weeks after intervention
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: percentage of apoB change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 468
percentage of apoB change | 2.42 (50.48)

8. Secondary Outcome: Change in Serum Alanine Aminotransferase
Description: Blood tests
Time Frame: Baseline up to 8 weeks after intervention
Population: Safety set
Measure: Median (Full Range); unit: percentage of ALT change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 492
percentage of ALT change | 0.00 [-72.92 to 1118.75]

9. Secondary Outcome: Change in Serum Aspartate Aminotransferase
Description: Blood tests
Time Frame: Baseline up to 8 weeks after intervention
Population: Safety set
Measure: Median (Full Range); unit: percentage of AST change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 492
percentage of AST change | 10.91 [-77.73 to 676.47]

10. Secondary Outcome: Change in Serum Creatine Kinase
Description: Blood tests
Time Frame: Baseline up to 8 weeks after intervention
Population: Safety set
Measure: Median (Full Range); unit: percentage of CK change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 492
percentage of CK change | 8.02 [-73.94 to 1429.63]

11. Secondary Outcome: Change in Serum Creatinine
Description: Blood tests
Time Frame: Baseline up to 8 weeks after intervention
Population: Safety set
Measure: Median (Full Range); unit: percentage of Creatinine change
Arm/Group | Fenofibrate Arm
Number analyzed (Participants) | 492
percentage of Creatinine change | 12.99 [-63.63 to 80.43]

12. Secondary Outcome: Change in Serum High Sensitivity C-reactive Protein
Description: Blood tests
Time Frame: Baseline and up to 8 weeks after intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks + 1 month
Description: Serious Adverse Events were collected after Informed Consent was signed.
Arm/Group | Fenofibrate Arm
Serious Adverse Events (participants affected / at risk) | 7/492
Other Adverse Events (participants affected / at risk) | 23/492
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate Arm (N=492)
Hepatic enzyme increased (Hepatobiliary disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate Arm (N=492)
Nausea (Gastrointestinal disorders) | 5 (5)
Alanine aminotransferase increased (Investigations) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 6 (6)
Blood creatine phosphokinase increased (Investigations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other